CLINICAL TRIAL: NCT01343719
Title: A Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Phase I Study to a) Assess Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of 2 mg to 350 mg of BI 661051 Administered as Oral Drinking Solution (Powder in Bottle) in Healthy Male Volunteers, b) to Explore the Relative Oral Bioavailability of a Tablet Formulation and c) to Assess the Impact of a High Fat Meal on the Oral Bioavailability of the Oral Drinking Solution (Powder in Bottle)
Brief Title: Single Rising Dose Study to Assess Safety, Tolerability and Pharmacokinetics of BI 661051.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1296.1; 2010-022465-96 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-19; First posted 2011-04-28 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (11):
- BI 661051 low dose, low (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 low dose, medium (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 low dose, high (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 medium dose, low (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 medium dose, medium (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 medium dose, high (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 high dose, low (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 high dose, medium (Experimental): solution for oral administration, single dose
  Interventions: Drug: BI 661051
- BI 661051 low dose (Experimental): tablet
  Interventions: Drug: BI 661051
- BI 661051 medium dose (Experimental): tablet
  Interventions: Drug: BI 661051
- Placebo (Placebo Comparator): solution for oral administratrion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 661051 — medium dose solution for oral administration
  Arms: BI 661051 medium dose, low
Drug: BI 661051 — medium dose solution for oral administration
  Arms: BI 661051 medium dose, medium
Drug: BI 661051 — medium dose solution for oral administration
  Arms: BI 661051 medium dose, high
Drug: BI 661051 — low dose solution for oral administration
  Arms: BI 661051 low dose, high
Drug: BI 661051 — low dose solution for oral administration
  Arms: BI 661051 low dose, low
Drug: BI 661051 — low dose solution for oral administration
  Arms: BI 661051 low dose, medium
Drug: BI 661051 — high dose solution for oral administration
  Arms: BI 661051 high dose, low
Drug: BI 661051 — high dose solution for oral administration
  Arms: BI 661051 high dose, medium
Drug: BI 661051 — low dose tablet
  Arms: BI 661051 low dose
Drug: Placebo — solution for administration
  Arms: Placebo
Drug: BI 661051 — medium dose tablet
  Arms: BI 661051 medium dose

SUMMARY:
The objective of the current study is to investigate safety, tolerability, and pharmacokinetics of treatment with BI 661051 rising single doses administered as oral drinking solution (powder in bottle) in healthy male subjects.

The primary objective is to investigate the safety and tolerability of treatment with BI 661051.

The secondary objectives are (1) to evaluate the single dose pharmacokinetics of BI 661051, (2) to explore dose proportionality, (3) to explore the relative bioavailability when BI 661051 is administered as tablet at two dose levels compared to oral drinking solution and (4) to assess the effect on the bioavailability when BI 661051 is administered as oral drinking solution after intake of a high fat meal.

Pharmacodynamic parameters will not be determined within this study.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

1. Healthy males based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
2. Age =18 and age =50 years.
3. BMI =18.5 and BMI =30 kg/m2 (Body Mass Index).
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance.
2. Any evidence of a clinically relevant concomitant disease.
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders.
5. History of relevant orthostatic hypotension, fainting spells or blackouts.
6. Chronic or relevant acute infections.
7. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients) as judged clinically relevant by the investigator.
8. Intake of drugs with a long half-life (>24 h) within at least 1 month or less than 10 half-lives of the respective drug prior to administration.
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomisation.
10. Participation in another trial with an investigational drug within 30 days prior to randomisation.
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day).
12. Inability to refrain from smoking on trial days as judged by the investigator.
13. Alcohol abuse (more than 30 g/day).
14. Drug abuse.
15. Blood donation (more than 100 mL within 4 weeks prior to randomisation or during the trial).
16. Excessive physical activities (within 1 week prior to randomisation or during the trial).
17. Any laboratory value outside the reference range that is of clinical relevance.
18. Inability to comply with dietary regimen of the study centre.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of findings of physical examination | 14 weeks
Vital signs (blood pressure (BP), pulse rate (PR), respiratory rate [RR]) | 14 weeks
Orthostasis test parameters | 14 weeks
Body temperature | 14 weeks
12-lead electrocardiogram (ECG) parameters (heart rate, PQ interval, QRS interval, uncorrected QT interval as well as Bazett- and Fridericia corrected QT interval) | 14 weeks
Clinical laboratory test parameters (haematology, clinical chemistry and urinalysis parameters) | 14 weeks
Occurrence of adverse events (AEs) on the level of Medical Dictionary for Regulatory Affairs (MedDRA) Preferred Terms and MedDRA System Organ Class | 14 weeks
Occurrence of findings detected by the pupillometry measurements | 14 weeks
Tolerability assessed by investigator | 14 weeks

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | 14 weeks
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | 14 weeks
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable analyte plasma concentration) | 14 weeks
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1296.1.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany